# Evaluation of the analgesic efficacy of the combination of deksketoprofen + paracetamol and the combination of naproxen sodium + codeine in patients with acute dental pain

İbrahim Doğru<sup>1</sup>, Levent Ciğerim<sup>1</sup>

<sup>1</sup> Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery, Van,

## **TURKEY**

Corresponding author: İbrahim Doğru

Address: Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery,

Van, Turkey Postal Code: 65080

E-mail address: <u>ibrahimdogru@yyu.edu.tr</u> Phone:+905418952655 Office Phone: 904322251744 Fax:

+904322251747

#### İbrahim DOĞRU

Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery <a href="mailto:ibrahimdogru@yyu.edu.tr">ibrahimdogru@yyu.edu.tr</a>, +905418952655, <a href="https://orcid.org/0000-0001-9174-9401">https://orcid.org/0000-0001-9174-9401</a>

### Levent CİĞERİM

Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery <a href="mailto:leventcigerim@yyu.edu.tr">leventcigerim@yyu.edu.tr</a>, +905321633287, <a href="https://orcid.org/0000-0001-5218-8568">https://orcid.org/0000-0001-5218-8568</a>

## VAN YÜZÜNCÜ YIL UNIVERSITY DURSUN ODABAŞ MEDICAL CENTER INFORMED CONSENT FORM FOR RESEARCH

### Dear patient,

Please read this document carefully and listen carefully to what we have said. Detailed information about the research; Detailed information about your rights, benefits and risks of the research can be found in this document. The purpose of these statements is to inform you about your health. Please indicate what you do not understand, your questions will be explained in detail. You can leave the research at any stage of the research if you think that your questions are not adequately explained after you accept to participate in the research or for any other reason. During the research period, the health problems arising from our research will be treated in our hospital immediately. You will not be charged an additional fee for participating in this research, nor will you be paid. Thank you for participating in our research.

## Name of the research:

Evaluation of the analgesic efficacy of the combination of deksketoprofen + paracetamol and the combination of naproxen sodium + codeine in patients with acute dental pain

## Subject, purpose, method, duration and process of the research:

In our study, the drugs used for severe toothache caused by infection in impacted lower wisdom teeth usually include naproxen sodium + codeine phosphate, dexketoprofen trometamol + paracetamol. Our trial will compare the pain relief of these drugs.

People like you who have pain caused by a half-implanted wisdom tooth will start taking one of the medicines 7 days early. At the end of the 7 days, your opinion on the effectiveness of the painkiller will be asked and the effects of the drugs will be compared.

The method of our study: Our study is about the evaluation of the effectiveness of the painkiller that you will be given. In the evaluation of this efficacy, you will be given a form for pain assessment and you will be asked to fill in this form by scoring the level of pain you feel at the specified times for 7 days between 0 (no pain) and 10 (unbearable pain).

**The duration and process:** our research will end when you inform us about the pain relief effectiveness of the medication given to you within 7 days before the procedure and the tooth that causes pain is extracted.

A brief description of the proposed procedure/process related to the study: For 7 days you will be asked to take the medication and record pain scores and other drug effects. At the end of the 7th day, the procedure will end with the extraction of the tooth causing pain.

Possible harms or risks that the patient/volunteer may encounter during the research: Depends on the medicines used in the study: Allergy, nausea, vomiting, diarrhoea, gastrointestinal problems, fever, dizziness, headache, visual disturbances, cardiovascular problems, kidney/liver problems, loss of appetite, tinnitus, loss of attention, depression, addiction, anaemia, constipation, etc. Other possible medication side effects may occur. In this case, immediate medical attention will be provided by your doctor.

**Possible benefits of the study:** Our research will offer the following benefits to you/society: As a result of our research, the efficacy of the drugs we will use in patients will be evaluated and the most effective pain relief drug components for severe toothache will be determined and the current results will be presented to the public and the scientific world for evaluation. Thus, in the light of this information, the evaluation of the drugs to be used in the future will be healthier.

Study-specific risks that may occur during the study: Yes



No



Dear patient/ participant/....., please read the following articles carefully and fill in the relevant blank or tick the relevant box